CLINICAL TRIAL: NCT07076992
Title: The Dilemma of Neonatal Circumcision in Egypt: A Comparative Randomized Study
Brief Title: Dilemma of Neonatal Circumcision in Egypt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Ahmed Elmaadawy, Lecturer of Urology, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 36264PR1075/1/25
Record Dates: First submitted 2025-07-02; First posted 2025-07-22 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Neonate; Circumcision

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Patients will undergo circumcision by Plastibell (PB).
  Interventions: Procedure: Circumcision by Plastibell
- Group 2 (Experimental): Patients will undergo circumcision by the Gomco (GM).
  Interventions: Procedure: Circumcision by Gomco

INTERVENTIONS:
Procedure: Circumcision by Plastibell — Patients will undergo circumcision by Plastibell (PB).
  Arms: Group 1
Procedure: Circumcision by Gomco — Patients will undergo circumcision by the Gomco (GM).
  Arms: Group 2

SUMMARY:
The study aims to compare wound healing, wound healing complications, cosmetic outcome, and level of parental satisfaction amongst four techniques of neonatal circumcision.

DETAILED DESCRIPTION:
Circumcision of a male child is the most common surgery performed globally. The prevalence of circumcision in this part of the world is over 80%, with the majority conducted in the neonatal period. The techniques of circumcision are diverse, and the method of circumcision may account for the differences in the outcome of the procedure.

Circumcision has complications like all surgical procedures. These typically include early complications such as leakage, hemorrhage, wound infection, pain, and swelling. However, more serious problems such as prolonged bleeding and amputation of the glans penis may also be encountered.

ELIGIBILITY:
Inclusion Criteria:

* Male infants less than 3 months old.
* Undergoing circumcision.

Exclusion Criteria:

* Male infants more than 3 months old.
* Infants with bleeding disorders.
* Neonates with hypospadias, epispadias, micropenis, disorders of sex development (DSD)
* Neonates with buried or webbed penis.

Max Age: 3 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male infants undergoing circumcision
Enrollment: 60 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Post circumcision bleeding | 2 hours postoperatively
  All infants will be followed up for 2 hours for early detection and management of post circumcision bleeding.

SECONDARY OUTCOMES:
Wound healing | 7 days postoperatively
  Superficial wound healing will be assessed on the 7th post-operative day.
Parental satisfaction | 4 weeks postoperatively
  Degree of parental satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.